CLINICAL TRIAL: NCT04296617
Title: Assessment of Predicted LET and Dosimetry in Relation to White Matter Changes in Pediatric Patients Following Proton Therapy for Primary Central Nervous System and Base of Skull Malignancies: A Pilot Study
Brief Title: Brain Imaging Changes Following Proton Therapy for Pediatric Primary Central Nervous System and Base of Skull Tumors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1777; NCI-2020-01197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-002279 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Malignant Central Nervous System Neoplasm; Malignant Skull Base Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical chart review): Patients' medical charts are reviewed.
  Interventions: Other: Medical Chart Review

INTERVENTIONS:
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review

SUMMARY:
This trial gathers information from patients with primary central nervous system or base of skull tumors that receive proton beam therapy and see if certain imaging techniques can help detect radiation-related changes over time. This study may help providers learn more about proton beam radiotherapy and how to improve the way it is delivered.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish linear energy transfer (LET)-based models as early predictors for white matter changes on magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI) sequences in pediatric patients following proton beam therapy for primary central nervous system (CNS) and base of skull tumors.

OUTLINE:

Patients' medical charts are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed central nervous system of skull base tumors
* Patient is going to undergo central nervous system (CNS) or base of skull proton beam therapy

Exclusion Criteria:

* Patients who have received prior therapeutic radiotherapy to the primary brain tumor site
* Patients who are unable to maintain follow-up through the Phoenix Children's Hospital and Mayo Clinic Arizona

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are diagnosed with central nervous system or base of skull malignancies, undergoing proton beam therapy
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
White matter changes within the central nervous system (CNS) following proton beam therapy using magnetic resonance imaging (MRI) sequences | At 18 months
  The concordance of predicted linear energy transfer linear (LET) values with radiographic white matter changes will be analyzed utilizing a one sample t-test. Will the compare concordance over time to evaluate if there is an increase, utilizing repeated measures mixtures models.
White matter changes within the CNS following proton beam therapy using diffusion tensor imaging (DTI) sequences | At 18 months
  The concordance of predicted LET values with radiographic white matter changes will be analyzed utilizing a one sample t-test. We will the compare concordance over time to evaluate if there is an increase, utilizing repeated measures mixtures models.
Relative biological effectiveness (RBE) predictions | Up to 18 months
  Will compare concordance over time to evaluate if there is an increase, utilizing repeated measures mixtures models.

SECONDARY OUTCOMES:
White matter changes within the CNS following proton beam therapy using DTI and MRI | Up to 18 months
  Will assess the white matter changes within the CNS following proton beam therapy using DTI and MRI and determine concordance with predicted RBE values and biological dose.
Dose-volume effect and predicted LET distribution | Up to 18 months
  Will be correlated. Will evaluate the percent of concordance of isodose volumes with white matter changes utilizing pairwise t-tests and repeated measures mixed models.
White matter changes identified on imaging, and predict concordance | Up to 18 months
  Will be described with both clinical acute and late toxicities following proton beam therapy. Exploratory analyses utilizing tests for association and appropriate regression techniques will be conducted to determine the association of dose volume histogram, LET, RBE, and clinical factors on acute and late toxicities caused by white matter changes.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Z. Vern-Gross, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials